CLINICAL TRIAL: NCT05087147
Title: Clinical Evaluation of Bonded Versus Banded Space Maintainers in Children With Prematurely Lost First Primary Molars: A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of Bonded Versus Banded Space Maintainers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Omar Sherif Ahmed Abo El Abbas (Other)
Responsible Party: Sponsor-Investigator, Omar Sherif Ahmed Abo El Abbas, Assistant Lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: space maintainer
Record Dates: First submitted 2021-09-27; First posted 2021-10-21 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Masking Description: Statisticians
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bonded space maintainer (Experimental): Wire bonded with composite to abutment teeth
  Interventions: Device: 0.7 mm stainless steel orthodontic wire
- Banded space maintainer (Active Comparator): Band and loop space maintainer
  Interventions: Device: Banded space maintainer

INTERVENTIONS:
Device: 0.7 mm stainless steel orthodontic wire — 0.7 mm stainless steel orthodontic wire
  Arms: Bonded space maintainer
Device: Banded space maintainer — band and loop space maintainer
  Arms: Banded space maintainer

SUMMARY:
Comparing bonded space maintainers to banded space maintainers

DETAILED DESCRIPTION:
Comparing bonded space maintainers to banded ones regarding clinical success in maintaining the space for the prematurely lost primary molar and radiographic space loss in both banded and bonded space maintainers. Finally, patient satisfaction regarding both treatments.

ELIGIBILITY:
Inclusion criteria:

Patient and parent showing cooperation and compliance. Medically free children. Patients having mandibular first deciduous molar indicated for extraction due to extensive coronal caries beyond possible repair, root caries and/or failed pulp therapy.

Having all first permanent molars erupted and in Class I molar relation. According to space analysis available space is less than or equal to needed space.

Having all their mandibular incisors erupted. With deciduous canines and second deciduous molars in the side of the extraction maintained throughout the entire follow-up period. Caries free, non-restored buccal surfaces of the mandibular second primary molars and deciduous canines. 1/3 to less than 2/3 of the root of the permanent successor is formed to the prematurely lost primary molars.

Exclusion criteria:

Children with any parafunctional habits. Children with previous allergies to stainless steel. Crowned abutment teeth. Permanent successors with 2/3 of its roots formed and space analysis does not indicate the fabrication of space maintainer.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
appliance failure | up to 12 months
  Patient reported

SECONDARY OUTCOMES:
Radiographic space loss | up to 12 months
  in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Omar S Abo El Abbas, Principal Investigator — Cairo U

IPD SHARING:
Plan to Share IPD: No